CLINICAL TRIAL: NCT06380738
Title: A Prospective Observational Study to Evaluate Real-world Clinical Outcomes and Characteristics of Patients With mCRPC Treated With Olaparib + Abiraterone
Brief Title: Real-World Clinical Experience of Patients With Metastatic Castration-Resistant Prostate Cancer Treated With Olaparib + Abiraterone (PROceed)
Acronym: PROceed
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: D0817R00074; D0817R00074 (Other: AstraZeneca)
Record Dates: First submitted 2024-02-01; First posted 2024-04-24 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Castration-resistant Prostate Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
PROceed is a multisite, prospective, observational study that describes the real-world use and clinical experience of mCRPC patients treated with the combination of olaparib and abiraterone in the mCRPC setting. Clinical outcomes will be assessed in patients who are either NHA-naive or NHA-exposed prior to initiating olaparib + abiraterone treatment, respectively. Patient demographic and clinical characteristics, as well as treatment received prior and subsequent to olaparib + abiraterone, will also be described. The study plans to enroll patients for a maximum of 2 years and follow up patients from initiation of olaparib until 1 year post last patient in.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent;
* 18 years of age and above;
* Documented histopathology or cytopathology of PCa, adenocarcinoma;
* Confirmed as mCRPC;
* Initiated olaparib + abiraterone after site activation

Exclusion Criteria:

* Patients participating in a clinical trial with an investigational prostate cancer treatment within 30 days prior to olaparib initiation

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of patients with a confirmed mCRPC diagnosis that has initiated the combination of olaparib and abiraterone through routine clinical practice at participating sites in Germany.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-02-14 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Time to treatment discontinuation | Up to 12 months
  Time to treatment discontinuation (TTD) event-free rate at 6 months and 12 months will be assessed among patients treated with olaparib + abiraterone in 1L mCRPC setting by prior NHA exposure status (NHA-exposed and NHA-naive), respectively.
  TTD is defined as the time from initiation of olaparib therapy until end date of olaparib therapy or death due to any cause.

SECONDARY OUTCOMES:
Time to first subsequent therapy | Up to 24 months
  Time to first subsequent therapy (TFST) in mCRPC patients treated with olaparib + abiraterone.
  TFST is defined as the time from olaparib initiation to the earlier of the first subsequent anticancer therapy start date following olaparib discontinuation or death due to any cause.

CONTACTS AND LOCATIONS:
Locations (34):
- Germany (34):
  - Research Site, Aschaffenburg
  - Research Site, Augsburg
  - Research Site, Bergisch Gladbach
  - Research Site, Berlin
  - Research Site, Bonn
  - Research Site, Cologne
  - Research Site, Dresden
  - Research Site, Duisburg
  - Research Site, Eisenach
  - Research Site, Eisleben Lutherstadt
  - Research Site, Frankfurt
  - Research Site, Greifswald
  - Research Site, Halle
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Heidelberg
  - Research Site, Heinsberg
  - Research Site, Herzogenaurach
  - Research Site, Leipzig
  - Research Site, Lübeck
  - Research Site, Lüneburg
  - Research Site, Magdeburg
  - Research Site, Marburg
  - Research Site, Mülheim
  - Research Site, Münster
  - Research Site, Neunkirchen
  - Research Site, Nuremberg
  - Research Site, Rüsselsheim am Main
  - Research Site, Saalfeld
  - Research Site, Speyer
  - Research Site, Trier
  - Research Site, Tübingen
  - Research Site, Westerstede
  - Research Site, Wetzlar

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal
  Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/